CLINICAL TRIAL: NCT04441151
Title: Evaluation of the Effect of Pulmonary Rehabilitation on Patients With High Flow Oxygen Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Ph.D., Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pulmonary rehabilitation
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Pulmonary rehabilitation therapy
  Interventions: Behavioral: Pulmonary rehabilitation therapy
- Control group (No Intervention): Routine medical treatment

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation therapy — Comprehensive interventions based on comprehensive evaluation and customization of patients, including, but not limited to, exercise training, education and behavioral changes, aimed at improving the physiological and psychological status of patients with chronic respiratory diseases, and urge patients to adhere to health promotion activities for a long time.
  Arms: Experimental group

SUMMARY:
Evaluation of the effect of pulmonary rehabilitation on patients with high flow oxygen therapy

DETAILED DESCRIPTION:
Objective: the purpose of this study was to evaluate the effect of lung rehabilitation on patients treated with high flow humidification apparatus in ICU. Methods: 70 patients in ICU who were treated with high flow humidification apparatus from June 2019 to June 2020 were randomly divided into two groups. The experimental group was treated with pulmonary rehabilitation and the control group was treated with routine medical treatment only. All patients were evaluated and measured by bedside diaphragm ultrasound. The vital signs of all patients were monitored every day. MRCsum assessment of peripheral muscle strength, 30s sitting test, modified Barthel index, Borg dyspnea score, arterial blood gas analysis and bedside diaphragm ultrasound monitoring were performed at admission and discharge. Finally, statistics were made on the use of non-invasive ventilator, endotracheal intubation, new complications (pressure sore, aspiration, thrombus, etc.) and the time of patients getting out of bed for the first time.The end point of the experiment was 28 days.

ELIGIBILITY:
Inclusion Criteria:

* The age is ≥ 18 years old;
* the hemodynamics is stable;
* 50 < heart rate < 120 beats / min ;
* 90 < systolic blood pressure < 200mmHg ;
* 55 < mean arterial pressure < 120mmHg;
* do not increase the dose of pressor drugs for at least 2 hours;
* intracranial pressure is stable and there are no seizures within 24 hours;
* the respiratory state is stable;
* the patient's finger pulse oxygen saturation ≥ 88%;
* 10 < respiratory frequency < 35 beats / min.

Exclusion Criteria:

* Pregnancy;
* acute cardio-cerebrovascular events;
* spinal or limb fractures;
* active bleeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
MRC | Day 28
  Medical Research Council,Muscle strength assessment,total points0~60，less than 48scores means ICU aquired weaknesses.
STS | Day 28
  Number of sit-to-stand test in 30s,Muscle endurance assessment,The more times, has the better muscular endurance.
barthel index | Day 28
  barthel index,Daily activity assessment,Assessment of activities of daily living.total points0~100，less than 60 scores means can't independent living.
Borg dyspnea score | Day 28
  Borg dyspnea score,Maximum 10 points,Minimum 0,The higher the score, the harder it is to breathe
PaO2 | Day 28
  arterial partial pressure of oxygen,Partial pressure of oxygen in arterial blood,normal range is 80~100.
Oxygenation index | Day 28
  arterial partial pressure of oxygen divided by the oxygen concentration,Normal is greater than 400.
Diaphragm mobility | Day 28
  The distance the diaphragm drops during inhalation,normal is 1.4cm.
Diaphragm contraction velocity | Day 28
  The rate at which the diaphragm contracts during inhalation,normal is 1.3cm/s.
End-inspiratory diaphragm thickness | Day 28
  The thickness of the diaphragm during inhalation,The thickness of diaphragm at the end of expiratory is about 0.25cm.
End-expiratory diaphragm thickness | Day 28
  The thickness of the diaphragm during exhalation,The thickness of diaphragm at the end of expiratory is about 0.15cm.
Diaphragm thickness variation rate | Day 28
  Rate of diaphragmatic thickness change during breathing,Diaphragmatic dysfunction is considered less than 20%.

SECONDARY OUTCOMES:
ICU stay time | 3 month
  icu length of stay
Hospitalization time | Month 3
  Hospitalization time,length of stay in hospital.
The time it takes to get out of bed for the first time | Day 28
  The time it takes to get out of bed for the first time
Use of non-invasive ventilator | Day 28
  Use of non-invasive ventilator,Whether to use non-invasive ventilator within 28 days.
Intubation | Day 28
  Intubation,Whether endotracheal intubation was performed for invasive mechanical ventilation within 28 days
mortality | Day 28
  mortality
Complication | Day 28
  The incidence of new complications(pressure sores、thrombus、aspiration).

CONTACTS AND LOCATIONS:
Overall Officials: wang, doctor, Principal Investigator — The First Medical Center of PLA General Hospital
Locations (1):
- Chinese PLAGH Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No